CLINICAL TRIAL: NCT03059342
Title: Short and Longterm Evolution of Self-care and Functional Mobility After Single Event Multilevel Surgery in Children and Adolescents With Spastic Diplegic Cerebral Palsy
Brief Title: Functional Follow-up After Single Event Multilevel Surgery in Children Spastic Diplegic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Griet Dequeker, MSC Occupational Science, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S54835
Record Dates: First submitted 2017-02-02; First posted 2017-02-23 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Cerebral Palsy
Keywords: spastic diplegic CP; self-care; functional mobility; multilevel surgery
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: single event multilevel surgery

SUMMARY:
Purpose: The aim of this study is to assess the short- and midterm evolution of self-care and functional mobility after multilevel surgery in children and adolescents with spastic diplegic cerebral palsy and to identify which factors could have an impact on these outcomes.

Methods: Thirty-four participants were included. All participants will be evaluated before surgery, at 9 weeks, 6,12,18, 24, 36 and 60 months. Self-care was assessed with the Pediatric Evaluation of Disability Inventory-NL (PEDI-NL). The Mobility Questionnaire47 (MobQues47) and Functional Mobility Scale (FMS) were used to measure functional mobility. Interactions between CP, personal and environmental characteristics and evolution in time were assessed.

DETAILED DESCRIPTION:
1. Introduction Cerebral palsy (CP) is the most common physical disability with a prevalence between two and three per 1000 living births. Cerebral palsy had been defined as a group of permanent disorders of the development of movement and posture, causing activity limitations that are contributed to non-progressive disturbances that occurred in the developing fetal and infant brain. The motor disorders are often accompanied by disturbances of sensation, perception, cognition, communication and behavior, by epilepsy and by secondary musculoskeletal problems. Cerebral palsy can have an impact on the body function and on the performance of daily life activities and as such may affect the child's independence, participation and quality of life.

The impact of cerebral palsy on individuals varies widely. The SCPE describes a hierarchical classification tree of cerebral palsy subtypes: spastic CP, dyskinetic CP and ataxic CP. Spastic CP is the most common type and is seen in 85% of the children with CP. The Gross Motor Function Classification System (GMFCS) classifies children and adolescents with cerebral palsy in five levels on the basis of their functional abilities in sitting and walking. Further subdivision is made according to the topographical distribution i.e. hemiplegia, diplegia and quadriplegia. Howard et al. reported that in a group of 323 children with spastic cerebral palsy 35 % of children had hemiplegia, 28 % diplegia and 37% quadriplegia. In their study the GMFCS levels of spastic diplegic cerebral palsy were 33% with GMFCS I, 33 % GMFCS II, 28% GMFCS III and 5% GMFCS IV. This means that nearly all spastic diplegic patients have the ability to walk with or without assistive devices.

A multidisciplinary follow-up is necessary during growth of the child with CP. A good knowledge of normal developmental milestones and natural history of children with CP is important to detect and prevent early problematic situations. In normal development the period of early childhood is characterized by rapid development of locomotor skills as walking, running and stair climbing. Typically developing children learn the skill of walking between the ages of eight and eighteen months. Children further learn to talk, start potty training and start to develop their independence in self-care skills. Achieving independence in dressing may take up to four years. Tying shoelaces and completing all clothing fasteners is achieved at age of six years. During this time, parents gradually perform fewer of the tasks, and encourage their children to do more, with the ultimate goal of independence.

In comparison with typically developing children, a child with spastic diplegic CP will show delay in all milestones but will generally stand at eighteen months and most will walk independently by four years. In the self-care domain, over half of the children with cerebral palsy needed help or supervision in the areas of grooming, bathing, dressing, and toileting. The gross motor function and function of self-care skills is steadily improving. At the age of nine years most children with spastic diplegic CP reached their maximum functional potential. Öhrvall et al. described that many children with CP achieve independence but at a later age than typically developing children. They reported that children with high functioning levels in GMFCS and in the Manual Ability Classification System (MACS) could achieve good functional performance for self-care and mobility at the age of 12 years. For children with GMFCS and MACS level III and more only minor development of functional skills is seen with age, although task-orientated and goal-directed therapy can improve their functioning.

Despite the improvement in self-care with age, several studies reported that the gait pattern in children with CP is deteriorating. Due to increased muscle tone and weakness children with spastic diplegic CP walk with hip and knee flexion, inward rotation and toe walking, hereby secondary problems like muscle contractures and bony deformities slowly arise. Further during the adolescents year's rapid growth and increase of body weight can lead to worsening deformities and changes in ratio of body mass to strength. Decrease of this ratio has a negative effect on the gait pattern.

Orthopedic surgery aims to counteract the effect of natural history by preventing the deterioration and as such maintaining function and keeping the child ambulant. Instead of performing several single level surgeries during childhood - the birthday syndrome approach - the modern approach aims to correct both muscle imbalance and bone deformity at the same time. The latter approach is called single event multilevel surgery (SEMLS) and ensures only one admission to the hospital with one rehabilitation period. SEMLS is not a uniform procedure but is tailored to the child's needs by lengthening shortened muscle-tendon units and realigning bony levers. In the University Hospital of Pellenberg, botulinum toxin is frequently applied simultaneously to reduce spasticity. Botox treatment and surgical treatment must be seen as complementary rather than exclusive. They both deliver benefits to a more normal alignment and make optimal rehabilitation possible. In addition successful outcome after multilevel surgery requires intensive training for at least one year following surgery. Important rehabilitation goals are improvement of the range of motion, strength, balance and function.

Several studies have investigated the effects of SEMLS. Two studies identified the loss of muscle strength post SEMLS. Seniorou et al. reported that muscle strength did not reach pre-operative status one year after SEMLS. It has been shown that multilevel surgery corrects musculoskeletal pathology and significantly improves the gait pattern. In the study of Thomason et al. these results were maintained at five years after surgery. However an important goal for children and parents is not only to achieve a better gait pattern but also to obtained an improved functionality in daily life. Mc Ginley et al. and Graham et al. stressed the importance for more longterm studies with multidimensional outcome measures in all domains of the International Classification of Functioning, Disability and Health (ICF).

There is a lack of studies focusing on the impact of SEMLS on activity level like self-care and functional mobility. Still information on these outcomes is very important for children and parents before undertaken this intervention. After SEMLS the intensive rehabilitation period requires high physical and mental demands and the long lasting rehabilitation process could be strenuous for children and parents. Insufficient information about the post-surgery period could lead to frustration of the parents and children.

A few longitudinal studies measured functional mobility in daily life activities after SEMLS using the Functional Mobility Scale (FMS). Harvey et al.reported for a group of 66 children with spastic diplegic CP a deterioration at three and six months post-surgery, followed by improvement back to baseline status at one year and further improvement at two years post-surgery. Another study in nine children with spastic diplegic CP showed one year after SEMLS no differences in the FMS. Children in this study underwent also bony foot surgery as part of SEMLS. In the follow-up study of Thomason et al. nearly half of the children had improved on the distance of 50 and 500 m five years post-surgery. In this study in 19 children with spastic diplegic CP no child deteriorated on the three distances of the FMS.

Only two studies reported effects of SEMLS in the domain of self-care skills. Buckon et al. compared the evolution of self-care after selective dorsal rhizotomy (SDR) and SEMLS using the PEDI in 25 children with spastic diplegia (18 SDR, 7 SEMLS). The SDR group showed significant gains for self-care skills at six months, one year and two years. The SEMLS group demonstrated no gains six months post-surgery. However at one and two year post SEMLS a significant increase in self-care skills was found. For the caregiver assistance only at two years post-surgery there was a significant decrease in the amount of assistance. Another study of Gorton et al. in 75 children with spastic CP (GMFCS I to III) reported no significant gain in scores on the Pediatric Functional Independence Measure (WeeFIM) one year post SEMLS.

Also some studies used Quality of life (QOL) measures after SEMLS. Two studies reported improvement of functional well-being one or two years after SEMLS. However the psychosocial and emotional wellbeing remained unchanged. Weak relationship between function and psychosocial domains of QOL was previously reported by Shelly et al. The study of Himpens et al. using the CP QOL showed that children with CP after SEMLS reported a higher quality of life compared to their parents reporting.

In summary, only a paucity of studies have been set up to study the effects on outcomes such as gross motor functional skills, activities of daily living functional skills and quality of life. Nevertheless it is necessary to examine the patient not only in gait laboratories but also in the context of daily life. Previous studies had only a short follow-up. There were based on a small sample size or had children with different types of CP . Further study is clearly needed to provide more insights in the short- mid- and longterm evolution of self-care and functional mobility following SEMLS.

Furthermore, knowledge of the factors influencing this evolution is of particular interest. Several CP related, personal and environmental characteristics may determine the evolution following surgery. The understanding of the associations between functional outcomes after SEMLS and potential influencing factors will aid to set realistic expectations and appropriate treatment plans after SEMLS. However, information on influencing factors on outcome of SEMLS is very limited. Svehlik et al. found better results following SEMLS for older children than younger children. The authors hypothesized that the finished growth spurt and probable better cooperation in therapy for the older children may lead to better outcomes. As Hoffinger indicated these results should be interpreted cautiously. Both groups in the retrospective study of Svehlik et al. are not the same. The older children had a poorer ambulation caused by primarily bone deformities, while the younger children had muscle contractures and muscle activation problems. Another study of Zwick et al. suggests that girls have better outcomes than boys. To date, only limited personal characteristics like age and gender were investigated as influencing factors, other possible interfering factors like GMFCS en MACS level, number of surgery and initial level on self-care and functional mobility have to be taken into account.

The aims of this study were to investigate the evolution in self-care and functional mobility at different time points over the first year following SEMLS and to assess if determinants could be identified that have an influence on these time trends.

Methods:

This prospective longitudinal study has a 5 year follow-up period. This study reports the short-term, midterm and longterm outcomes, i.e. at 2, 6, 12, 24, 36 and 60 months after SEMLS. Outcome measures were collected before surgery (time interval between one month to one day before surgery; T1) and at defined intervals after surgery, at 9 weeks (T2), 6 months (T3), 1 year (T4), 18 months (T5), 2 years (T6), 3 years (T7) and 5 years (T8). At this moment participants completed follow-up at 2 years.

All 34 participants were followed by the CP-reference center of the University Hospital of Pellenberg. The surgical recommendation was based to the participants' needs and determined by a comprehensive evaluation, including a standardized physical examination, radiographic evaluation and instrumental gait analysis.

All children and adolescents were hospitalized for one week after surgery in the University Hospital of Pellenberg. One week post-surgery they were discharged wearing plaster casts below-the-knee and removable knee braces. Participants received physiotherapy at home (five times a week) which consisted of passive joint mobilization. Four weeks after surgery participants were hospitalized again for rehabilitation at the University Hospital of Pellenberg or at the rehabilitation center 'Pulderbos' at Zandhoven. Rehabilitation comprised intensive individualized physiotherapy including an exercise programme of two hours per day, two hours positioning (standing table and specific stretch positions in prone and supine). The exercise programme consists of strength training and gait reeducation. Additionally, occupational therapy was provided if necessary (three times a week, 30-45 minutes) and focused on training upper limb function, transfers and activities of daily living (eating, washing, grooming,…). The rehabilitation period (hospital Pellenberg or rehab center Pulderbos) ranged from six to twelve weeks. Children and adolescents were discharged from the rehabilitation unit when independent walking with kaye-walker was possible. At home, rehabilitation was continued with the private physiotherapist with a frequency of five times a week up to six months post-surgery. At six months the frequency was individually adopted according to their needs. The children attending special education school had physiotherapy at school combined with private physiotherapy. The rehabilitation programme was similar in the two involved centres.

The Pediatric Evaluation of Disability Inventory (PEDI), Mobility Questionnaire47 (MobQues47), Functional Mobility Scale (FMS) and Manual Muscle Testing (MMT) were measured before surgery and after surgery at nine weeks, six months and one year. The CP QOl Child was measured before SEMLS and at one, three and five years following surgery.

All baseline assessments were conducted in the hospital of Pellenberg, assessment at nine weeks after surgery was performed at the rehabilitation unit, i.e. Pellenberg or Pulderbos. The following assessments took place during the follow-up consultations in the University Hospital of Pellenberg. The same assessor (senior occupational therapist) evaluated all participants, supported by two junior physiotherapists. Clinical assessments were practiced jointly in order to standardize assessment procedures.

Age, gender, intelligence and type of school, the level of Gross Motor Function Classification System (GMFCS) and Manual Ability Classification System (MACS) were collected before surgery. Also the surgical procedures and botulinum injections were documented.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of diplegic CP (Rosenbaum et al., 2007);
* GMFCS levels I, II, and III;
* aged between 6 and 25 years;
* bilateral surgery.

Exclusion Criteria:

* other diagnosis than cerebral palsy;
* severe mental retardation (IQ < 50).

Ages: 6 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: All consecutive children and adolescents with spastic diplegic CP who underwent multilevel surgery in the University Hospital of Pellenberg were screened for entry in the study between December 2012 and August 2014. SEMLS was defined as orthopedic surgery (soft-tissue or bony surgical procedures, combined or not with botulinum toxin injection) at two or more anatomical levels during one operative procedure, requiring only one hospital admission and rehabilitation period.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2012-12-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
change from baseline in self-care with the PEDI | after 9 weeks, 6,12,18,24,36 and 60 months
  The domain of self-care was evaluated by the Pediatric Evaluation of Disability Inventory (PEDI) (Haley, 1992). In this study, the functional skills and caregiver assistance for the domain of self-care were assessed by interview of the parent. For the domain self-care the PEDI-FSS measures skill mastery on 74 items (0 unable, 1 capable) whereas the PEDI-CAS measures the amount of assistance provided during the daily performance of these functional skills on a 6-point ordinal point system (0 complete assistance, 5 independent). Scores were calculated and transformed to interval-scaled scores (0-100), where 0 represents no ability and 100 indicates full capability. The Dutch version (PEDI-NL) (Wassenberg-Severijnen & Custers, 2005) was used. Several studies showed good reliability and excellent discriminative validity for the population of CP for the PEDI-NL (Custers et al., 2002; Wassenberg-Severijnen et al., 2003).
change from baseline in functional mobility with the Functional Mobility Scale | after 9 weeks, 6,12,18,24,36 and 60 months
  the Functional Mobility Scale (FMS) (Harvey, Graham, Morris, Baker, & Wolfe, 2007) The FMS rates the mobility of children with CP on a 6-point ordinal scale based on the need for assistive devices at three specific distances: 5, 50 and 500 m. These distances represent home, school and community environments respectively. The FMS is administered by asking a few questions on the child/parent. The scale is reliable and valid and has been able to detect changes after SEMLS (Harvey et al., 2007).
change from baseline in functional mobility with the Mobility Questionnaire47 | after 9 weeks, 6,12,18,24,36 and 60 months
  The Mobility Questionnaire (MobQues47, Van Ravesteyn, Dallmeijer, Scholtes, Roorda, & Becher, 2009) The Dutch version of the Mobility Questionnaire (MobiliteitsVragenlijst) (Van Ravesteyn et al., 2010a) was used. This questionnaire consists of 47 items like standing and walking on bare feet, stepping on and off a bike, going in and out of a car,… experienced by the children in their own home environment (with assistive devices if normally used). The mobility limitations were rated by the parents on a 5-point ordinal questionnaire (0 not possible, 4 no problem). The total score was converted to a scale of 0 to 100. Low scores represent severe limitations of mobility. The MobQues47 was specific developed for children with CP and has good reliability and validity (Van Ravesteyn et al., 2010a; Van Ravensteyn, Scholtes, Becher, Roorda, Verschuren, & Dallmeijer, 2010b).

SECONDARY OUTCOMES:
change from baseline in muscle strenght with the MMT | after 9 weeks, 6,12,18,24,36 and 60 months
  Muscle strength was assessed with manual muscle testing (MMT) according to the Medical Research Council (MRC) using a 10-point ordinal scale (0 contraction not palpable -10 movement against gravity with maximum resistance). Muscle strength was measured in eight muscle groups: hip flexors, extensors, abductors and adductors, knee flexors and extensors, ankle dorsal and plantar flexors. A total score for muscle strength was calculated (0-80). Although the MMT is generally used in clinical practice and research, the reliability in children with CP was only tested for the upper limbs (Klingels et al., 2010). To verify the reliability of the MMT for the lower limbs, an inter-rater reliability study was performed for the purpose of this study. A standardized test procedure used in the Clinical Motion Analysis Laboratory of the University Hospital of Pellenberg was used.
quality of life with the CP Qol | before surgery, after 1,3 and 5 years
  Quality of life was measured with the Quality of life Questionnaire for children and teenagers with CP (CP QOl) (Waters et al., 2007). The Dutch version of the CP QOl-Child was used (Smits-Engelsman et al., 2008). It contains a parent/proxy report and a child self-report. Both for the original version of the CP QOL and the Dutch version, good reliability was established (Smits-Engelsman et al., 2008). The scale consists 66 items and contains six domains (social wellbeing and acceptance, participation and physical health, functioning, emotional wellbeing, family health and access to services). All questions are scored on a 9-point rating scale in which a score of 1 indicates very unhappy, and a score 9 very happy. For the domains of pain and impact of disability, a score of 1 indicates no pain, not concerned at all while a score of 9 refers to a lot of pain, very concerned. For each domain, total scores are calculated ranging from 0 to 100. Low scores represents a low quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Molenaers, PHD, Principal Investigator — UZ Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Surveillance of Cerebral Palsy in Europe. Surveillance of cerebral palsy in Europe: a collaboration of cerebral palsy surveys and registers. Surveillance of Cerebral Palsy in Europe (SCPE). Dev Med Child Neurol. 2000 Dec;42(12):816-24. doi: 10.1017/s0012162200001511. PMID 11132255
- [Background] Prevalence and characteristics of children with cerebral palsy in Europe. Dev Med Child Neurol. 2002 Sep;44(9):633-40. PMID 12227618
- [Background] Palisano RJ, Rosenbaum P, Bartlett D, Livingston MH. Content validity of the expanded and revised Gross Motor Function Classification System. Dev Med Child Neurol. 2008 Oct;50(10):744-50. doi: 10.1111/j.1469-8749.2008.03089.x. PMID 18834387
- [Background] Howard J, Soo B, Graham HK, Boyd RN, Reid S, Lanigan A, Wolfe R, Reddihough DS. Cerebral palsy in Victoria: motor types, topography and gross motor function. J Paediatr Child Health. 2005 Sep-Oct;41(9-10):479-83. doi: 10.1111/j.1440-1754.2005.00687.x. PMID 16150063
- [Background] Bell KJ, Ounpuu S, DeLuca PA, Romness MJ. Natural progression of gait in children with cerebral palsy. J Pediatr Orthop. 2002 Sep-Oct;22(5):677-82. PMID 12198474
- [Background] Wong V, Chung B, Hui S, Fong A, Lau C, Law B, Lo K, Shum T, Wong R. Cerebral palsy: correlation of risk factors and functional performance using the Functional Independence Measure for Children (WeeFIM). J Child Neurol. 2004 Nov;19(11):887-93. doi: 10.1177/08830738040190110701. PMID 15658794
- [Background] Beckung E, Hagberg G, Uldall P, Cans C; Surveillance of Cerebral Palsy in Europe. Probability of walking in children with cerebral palsy in Europe. Pediatrics. 2008 Jan;121(1):e187-92. doi: 10.1542/peds.2007-0068. Epub 2007 Dec 10. PMID 18070932
- [Background] Ohrvall AM, Eliasson AC, Lowing K, Odman P, Krumlinde-Sundholm L. Self-care and mobility skills in children with cerebral palsy, related to their manual ability and gross motor function classifications. Dev Med Child Neurol. 2010 Nov;52(11):1048-55. doi: 10.1111/j.1469-8749.2010.03764.x. Epub 2010 Aug 16. PMID 20722662
- [Background] Eliasson AC, Krumlinde-Sundholm L, Rosblad B, Beckung E, Arner M, Ohrvall AM, Rosenbaum P. The Manual Ability Classification System (MACS) for children with cerebral palsy: scale development and evidence of validity and reliability. Dev Med Child Neurol. 2006 Jul;48(7):549-54. doi: 10.1017/S0012162206001162. PMID 16780622
- [Background] Bottos M, Feliciangeli A, Sciuto L, Gericke C, Vianello A. Functional status of adults with cerebral palsy and implications for treatment of children. Dev Med Child Neurol. 2001 Aug;43(8):516-28. doi: 10.1017/s0012162201000950. PMID 11508917
- [Background] Gough M, Eve LC, Robinson RO, Shortland AP. Short-term outcome of multilevel surgical intervention in spastic diplegic cerebral palsy compared with the natural history. Dev Med Child Neurol. 2004 Feb;46(2):91-7. doi: 10.1017/s0012162204000192. PMID 14974633
- [Background] Graham HK, Harvey A. Assessment of mobility after multi-level surgery for cerebral palsy. J Bone Joint Surg Br. 2007 Aug;89(8):993-4. doi: 10.1302/0301-620X.89B8.19446. PMID 17785733
- [Background] Akerstedt A, Risto O, Odman P, Oberg B. Evaluation of single event multilevel surgery and rehabilitation in children and youth with cerebral palsy--A 2-year follow-up study. Disabil Rehabil. 2010;32(7):530-9. doi: 10.3109/09638280903180171. PMID 20136471
- [Background] Aiona MD, Sussman MD. Treatment of spastic diplegia in patients with cerebral palsy: Part II. J Pediatr Orthop B. 2004 May;13(3):S13-38. doi: 10.1097/00009957-200405000-00016. PMID 15083127
- [Background] Molenaers G, Van Campenhout A, Fagard K, De Cat J, Desloovere K. The use of botulinum toxin A in children with cerebral palsy, with a focus on the lower limb. J Child Orthop. 2010 Jun;4(3):183-95. doi: 10.1007/s11832-010-0246-x. Epub 2010 Mar 18. PMID 21629371
- [Background] Seniorou M, Thompson N, Harrington M, Theologis T. Recovery of muscle strength following multi-level orthopaedic surgery in diplegic cerebral palsy. Gait Posture. 2007 Oct;26(4):475-81. doi: 10.1016/j.gaitpost.2007.07.008. Epub 2007 Sep 12. PMID 17855096
- [Background] Thomason P, Baker R, Dodd K, Taylor N, Selber P, Wolfe R, Graham HK. Single-event multilevel surgery in children with spastic diplegia: a pilot randomized controlled trial. J Bone Joint Surg Am. 2011 Mar 2;93(5):451-60. doi: 10.2106/JBJS.J.00410. PMID 21368077
- [Background] Thompson N, Stebbins J, Seniorou M, Wainwright AM, Newham DJ, Theologis TN. The use of minimally invasive techniques in multi-level surgery for children with cerebral palsy: preliminary results. J Bone Joint Surg Br. 2010 Oct;92(10):1442-8. doi: 10.1302/0301-620X.92B10.24307. PMID 20884985
- [Background] Damiano DL, Abel MF, Pannunzio M, Romano JP. Interrelationships of strength and gait before and after hamstrings lengthening. J Pediatr Orthop. 1999 May-Jun;19(3):352-8. PMID 10344319
- [Background] McGinley JL, Dobson F, Ganeshalingam R, Shore BJ, Rutz E, Graham HK. Single-event multilevel surgery for children with cerebral palsy: a systematic review. Dev Med Child Neurol. 2012 Feb;54(2):117-28. doi: 10.1111/j.1469-8749.2011.04143.x. Epub 2011 Nov 24. PMID 22111994
- [Background] Thomason P, Selber P, Graham HK. Single Event Multilevel Surgery in children with bilateral spastic cerebral palsy: a 5 year prospective cohort study. Gait Posture. 2013 Jan;37(1):23-8. doi: 10.1016/j.gaitpost.2012.05.022. Epub 2012 Jul 19. PMID 22818117
- [Background] Capjon H, Bjork IT. Ambulant children with spastic cerebral palsy and their parents' perceptions and expectations prior to multilevel surgery. Dev Neurorehabil. 2010;13(2):80-7. doi: 10.3109/17518420903373511. PMID 20222768
- [Background] Harvey A, Graham HK, Morris ME, Baker R, Wolfe R. The Functional Mobility Scale: ability to detect change following single event multilevel surgery. Dev Med Child Neurol. 2007 Aug;49(8):603-7. doi: 10.1111/j.1469-8749.2007.00603.x. PMID 17635206
- [Background] Hoiness PR, Capjon H, Lofterod B. Pain and rehabilitation problems after single-event multilevel surgery including bony foot surgery in cerebral palsy. A series of 7 children. Acta Orthop. 2014 Dec;85(6):646-51. doi: 10.3109/17453674.2014.960141. Epub 2014 Sep 5. PMID 25191930
- [Background] Buckon CE, Thomas SS, Piatt JH Jr, Aiona MD, Sussman MD. Selective dorsal rhizotomy versus orthopedic surgery: a multidimensional assessment of outcome efficacy. Arch Phys Med Rehabil. 2004 Mar;85(3):457-65. doi: 10.1016/j.apmr.2003.05.009. PMID 15031833
- [Background] Gorton GE 3rd, Abel MF, Oeffinger DJ, Bagley A, Rogers SP, Damiano D, Romness M, Tylkowski C. A prospective cohort study of the effects of lower extremity orthopaedic surgery on outcome measures in ambulatory children with cerebral palsy. J Pediatr Orthop. 2009 Dec;29(8):903-9. doi: 10.1097/BPO.0b013e3181c11c0c. PMID 19934707
- [Background] Cuomo AV, Gamradt SC, Kim CO, Pirpiris M, Gates PE, McCarthy JJ, Otsuka NY. Health-related quality of life outcomes improve after multilevel surgery in ambulatory children with cerebral palsy. J Pediatr Orthop. 2007 Sep;27(6):653-7. doi: 10.1097/BPO.0b013e3180dca147. PMID 17717466
- [Background] Shelly A, Davis E, Waters E, Mackinnon A, Reddihough D, Boyd R, Reid S, Graham HK. The relationship between quality of life and functioning for children with cerebral palsy. Dev Med Child Neurol. 2008 Mar;50(3):199-203. doi: 10.1111/j.1469-8749.2008.02031.x. Epub 2008 Jan 21. PMID 18215191
- [Background] Himpens E, Franki I, Geerts D, Tack R, Van der Looven R, Van den Broeck C. Quality of life in youngsters with cerebral palsy after single-event multilevel surgery. Eur J Paediatr Neurol. 2013 Jul;17(4):401-6. doi: 10.1016/j.ejpn.2013.02.001. Epub 2013 Mar 6. PMID 23481663
- [Background] Svehlik M, Steinwender G, Kraus T, Saraph V, Lehmann T, Linhart WE, Zwick EB. The influence of age at single-event multilevel surgery on outcome in children with cerebral palsy who walk with flexed knee gait. Dev Med Child Neurol. 2011 Aug;53(8):730-5. doi: 10.1111/j.1469-8749.2011.03995.x. Epub 2011 Jun 29. PMID 21711455
- [Background] Hoffinger S. The influence of age on timing of single-event multilevel surgery: are adolescents with cerebral palsy comparable to a younger cohort? Dev Med Child Neurol. 2011 Aug;53(8):678-9. doi: 10.1111/j.1469-8749.2011.04038.x. Epub 2011 Jun 27. No abstract available. PMID 21707609
- [Background] Zwick EB, Svehlik M, Kraus T, Steinwender G, Linhart WE. Does gender influence the long-term outcome of single-event multilevel surgery in spastic cerebral palsy? J Pediatr Orthop B. 2012 Sep;21(5):448-51. doi: 10.1097/BPB.0b013e32834d4daa. PMID 22027704